CLINICAL TRIAL: NCT02328833
Title: Controlled Study About Implementation of a Computerized Depression Guideline in Primary Care
Acronym: GPC-DEPc
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Corporacion Parc Tauli (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Hospital Clinic of Barcelona (Other); Institut Catala de Salut (Other Government)
Responsible Party: Principal Investigator, Diego J. Palao-VIdal, Mental Health Director, Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SM-CSPT-DP2014-01
Record Dates: First submitted 2014-12-29; First posted 2014-12-31 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Depression
Keywords: Depression; Clinical Practice Guideline; Implementation; Primary Care; Computerized Guideline
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Implementation of Guidelines (Experimental): Primary Care Centers where the experimental strategies of guidelines implementation will be done
  Interventions: Other: Experimental strategies of guidelines implementation
- No Active Implementation of Guidelines (No Intervention): Primary Care Centers where the experimental strategies of guidelines implementation not will be done

INTERVENTIONS:
Other: Experimental strategies of guidelines implementation — Experimental strategies of Depression Guidelines implementation in Primary Care Centers. The active process includes the establishment of local implementation teams, seminars, regular feedback and follow-up visits for four months.
  Arms: Active Implementation of Guidelines

SUMMARY:
The aim of this study is to evaluate the effects of an active multifactor implementation process of a Computerized Depression Guideline in Primary Care. The CPG-DEPc use use, the key outcomes and its maintenance over time in patients and professionals will be analyzed.

DETAILED DESCRIPTION:
The application of scientific evidence on major depression in clinical practice is complex. Many studies show that over 50% of depressed patients in primary care do not receive proper attention, or are ineffective or potentially harmful treatments. In general, the process of dissemination and implementation of Clinical Practice Guidelines (CPG) in printed version induce a minor improvement in clinical practice. The adaptation of the CPG of Major Depression in Adults (CPG-DEPC) in Catalonia (Spain), as a computerized integrated version, offers an extraordinary opportunity to improve outcomes in Primary Care. The integrated design allows precise access to help in the visit itself, to improve diagnosis validation process, the recommended treatment and facilitate monitoring and evaluation of suicide risk in depressed patients.

This study aims to evaluate the effects of an active multifactor implementation process of a Computerized Depression Guideline in Primary Care. The GPC-DEPc use, the key outcomes and its maintenance over time in patients and professionals will be analyzed.

A cluster randomized trial, multicenter study in ten Primary Care Centers in Barcelona, coordinated by the same Mental Health Service, will be done. In five of the Centers will be actively implemented the CPG-DEPc and the other five will proceed as usual process, as a reference. The active process includes the establishment of local implementation teams, seminars, regular feedback and follow-up visits for four months. The main outcome will be the rate of patients with possible depression treated in the analyzed period in which at least were used any of the instruments that the Guide recommended (to rule out or confirm the diagnosis, choose the optimal treatment or follow-up the clinical maintenance best options). Other professionals and patients secondary outcome measures will be analyzed (incidence of major depression registers, referrals to mental health specialists, use of recommended antidepressants and rates of patients in clinical remission). At the end of the study, the suicide and suicide attempts rate and the data about the direct and indirect health cost will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years.
* Diagnosis of major depression (F32. **,F33.** according to International Classification of Diseases-10)
* Attended in any of the 10 selected Primary Care Centers (from Barcelona, Spain)
* Patients with suspected depression in which the diagnosis is discarded using the Guide.

Exclusion Criteria:

* Patients with diagnosed or suspected major depression treated by professionals who have not given their consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The rate of patients in which the instruments from the Computerized Depression Guideline were used. | 4 months
  The rate of patients with possible depression treated in the analyzed period in which at least one of the instruments that the Guide recommended were used (to rule out or confirm the diagnosis, choose the optimal treatment or the best clinical follow-up option).
The rate of patients in which the instruments from the Computerized Depression Guideline were used. | 6 months
The rate of patients in which the instruments from the Computerized Depression Guideline were used. | 12 months
The rate of patients in which the instruments from the Computerized Depression Guideline were used. | 18 months

SECONDARY OUTCOMES:
Incidence of major depression patients registered in the electronical clinical record. | 6 months
  New major depression cases (F32.**; F33.**) registered in the electronical clinical record.
Incidence of major depression patients registered in the electronical clinical record. | 12 months
Incidence of major depression patients registered in the electronical clinical record. | 18 months
Rates of suicide and suicide attempts | 18 months
Total health cost of depression | 18 months
  Direct and indirect health cost of major depression patients registered in electronical clinical record
Total referrals to mental health specialists | 6 months
Total referrals to mental health specialists | 12 months
Total referrals to mental health specialists | 18 months
Use Rate of the recommended antidepressives for the guideline | 6 months
Use Rate of the recommended antidepressives for the guideline | 12 months
Use Rate of the recommended antidepressives for the guideline | 18 months
Rate of patients in clinical remission | 6 months
  The clinical remission of depression symptoms is defined by a Patient Health Questionnaire-9 (PHQ-9) Score of < 5 points
Rate of patients in clinical remission | 12 months
Rate of patients in clinical remission | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Diego J Palao, Principal Investigator — Corporacion Parc Taulí Sabadell, University Hospital (Barcelona, Spain)

REFERENCES:
- [Background] Trinanes Y, Atienza G, Louro-Gonzalez A, de-las-Heras-Linero E, Alvarez-Ariza M, Palao DJ. Development and impact of computerised decision support systems for clinical management of depression: A systematic review. Rev Psiquiatr Salud Ment. 2015 Jul-Sep;8(3):157-66. doi: 10.1016/j.rpsm.2014.10.004. Epub 2014 Dec 12. English, Spanish. PMID 25500093
- [Background] Fernandez A, Pinto-Meza A, Bellon JA, Roura-Poch P, Haro JM, Autonell J, Palao DJ, Penarrubia MT, Fernandez R, Blanco E, Luciano JV, Serrano-Blanco A. Is major depression adequately diagnosed and treated by general practitioners? Results from an epidemiological study. Gen Hosp Psychiatry. 2010 Mar-Apr;32(2):201-9. doi: 10.1016/j.genhosppsych.2009.11.015. Epub 2010 Jan 12. PMID 20302995
- [Background] Serrano-Blanco A, Palao DJ, Luciano JV, Pinto-Meza A, Lujan L, Fernandez A, Roura P, Bertsch J, Mercader M, Haro JM. Prevalence of mental disorders in primary care: results from the diagnosis and treatment of mental disorders in primary care study (DASMAP). Soc Psychiatry Psychiatr Epidemiol. 2010 Feb;45(2):201-10. doi: 10.1007/s00127-009-0056-y. Epub 2009 May 19. PMID 19452110
- [Background] Pamias Massana M, Crespo Palomo C, Gisbert Gelonch R, Palao Vidal DJ. [The social cost of depression in the city of Sabadell (Barcelona, Spain) (2007-2008)]. Gac Sanit. 2012 Mar-Apr;26(2):153-8. doi: 10.1016/j.gaceta.2011.07.019. Epub 2011 Nov 3. Spanish. PMID 22055213
- [Background] Weinmann S, Koesters M, Becker T. Effects of implementation of psychiatric guidelines on provider performance and patient outcome: systematic review. Acta Psychiatr Scand. 2007 Jun;115(6):420-33. doi: 10.1111/j.1600-0447.2007.01016.x. PMID 17498153
- [Background] Sonnenberg FA, Hagerty CG. Computer-interpretable clinical practice guidelines. Where are we and where are we going ? Yearb Med Inform. 2006:145-58. PMID 17051309
- See also: Clinical Practice Guideline for Depression in Adults Patients of the National Health Spanish System (2014) — http://portal.guiasalud.es/GPC/GPC_534_Depresion_Adulto_Avaliat_resum.pdf
- See also: Adaptation to the Catalan Health Model of the Clinical Practice Guideline for Depression in Adults Patients of the National Health Spanish System (2010) — http://aquas.gencat.cat/web/.content/minisite/aquas/publicacions/2010/pdf/adaptacio_gpc_depressio_aiaqs_2010ca.pdf